CLINICAL TRIAL: NCT04056195
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Dose Study to Evaluate the Efficacy and Safety of Oral SKI-O-703, SYK Inhibitor, in Patients With Persistent and Chronic Immune Thrombocytopenia (ITP)
Brief Title: Study of Oral SKI-O-703, SYK Inhibitor, in Patients With Persistent and Chronic Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSCO-P2101
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2023-07

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — cevidoplenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SKI-O-703 200 mg (Experimental): 2 capsules of 100 mg SKI-O-703 BID (twice a day) 12 hours apart + 2 capsules of placebo during 12 weeks
  Interventions: Drug: SKI-O-703; Drug: Placebo oral tablet
- SKI-O-703 400 mg (Experimental): 4 capsules of 100 mg SKI-O-703 + 0 capsules of placebo during 12 weeks
  Interventions: Drug: SKI-O-703
- Placebo (Placebo Comparator): 4 capsules of placebo during 12 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: SKI-O-703 — The SKI-O-703 capsules will contain 100 mg of drug substance.
  Arms: SKI-O-703 200 mg; SKI-O-703 400 mg
Drug: Placebo oral tablet — Placebo capsules are filled with microcrystalline cellulose.
  Arms: Placebo; SKI-O-703 200 mg

SUMMARY:
Study in patients with persistent and chronic Immune Thrombocytopenia (ITP), who have failed to respond or relapsed after prior therapy, with a platelet count <30,000/µL. Patient will be randomly assigned in 2 groups with two dose levels of SKI-O-703 200mg BID, 400 mg BID, and placebo; administered orally twice a day.

DETAILED DESCRIPTION:
This study will evaluate the efficacy, safety, tolerability,pharmacokinetics (PK), and pharmacodynamics (PD) of select (200 mg BID and 400 mg BID) doses of SKI-O-703 in persistent and chronic ITP patients who have failed to respond or relapsed after prior therapy, with a platelet count <30,000/µL. on 2 occasions at least 7 days apart with the confirmatory count on the first day of treatment.

subjects will participate in 3 treatment groups (24 subjects in each of the active treatment groups and 12 subjects in the placebo group). The total study duration will be 20 weeks per subject, which consists of up to 4 weeks of screening period, 12 weeks of treatment period, and 4 weeks of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary ITP (persistent or chronic)
* Failed to respond or relapsed after at least 1 prior therapy, with a platelet count of <30,000/µL on 2 occasions at least 7 days apart with the confirmatory count on the first day of treatment
* Adequate hematologic, hepatic, and renal function
* ECOG performance status of 0, 1, or 2
* Male and female subjects, the subject and their partners of childbearing potential agree to use medically acceptable methods of contraception during the study and for 6 months following discontinuation of study drug (excluding women who are not of childbearing potential and men who have been sterilized. Men who have been sterilized should be confirmed to have negative sperm count on 2 consecutive occasions.)
* Male subjects agree not to donate sperm for 90 days after the last dose of study drug
* Female subjects have negative pregnancy tests at Screening.

Exclusion Criteria:

* History of current, active malignancy requiring or likely to require chemotherapeutic or surgical treatment during the study, with the exception of non-melanoma skin cancer, carcinoma in situ of the cervix, and localized prostate cancer managed by active surveillance
* Transfusion with blood or blood products or plasmapheresis within 2 weeks before the first administration of study drug
* History of known inherited coagulopathy, or recent arterial or deep venous thrombosis within the preceding 6 months
* Change in corticosteroid or immunosuppressant dose within 2 weeks prior to Day 1
* Treatment with thrombopoietin receptor agonists within 2 weeks before Day 1
* Treatment with rituximab or splenectomy within the 8 weeks prior to Day 1
* Treatment with intravenous immunoglobulins (IVIGs) within 4 weeks prior to Day 1
* Acute infection requiring oral antibiotics within 2 weeks
* Infections requiring intravenous antibiotics or hospitalization within 3 months
* Positive test results at Screening for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus antibody or positive result for hepatitis B core antibody with a negative result for hepatitis B surface antigen
* Received live vaccine within 28 days prior to Day 1 or plan to receive one during the study
* History or presence of any gastrointestinal, hepatic, or renal disease or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Uncontrolled hypertension
* Subject had 12-lead electrocardiogram (ECG) findings of corrected QT interval by Fridericia formula (QTcF) > 450 msec (males) or > 470 msec (females), cardiac arrhythmias, or clinically significant cardiac or ECG abnormalities
* Subject received any investigational medication within 30 days or 5 half-lives - Concomitant use of any anticoagulants and platelet aggregation inhibiting drugs including aspirin (within 14 days of planned dosing through end of follow-up)
* Female subject who is currently pregnant or breastfeeding
* Prior treatment with a SYK inhibitor
* Planned surgery in the time frame of the dosing period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (4):
  - University of Southern California, 1441 Eastlake Ave., Los Angeles, California
  - Duke University Medical Center, 2301 Erwin Road, Durham, North Carolina
  - East Carolina University, 600 Moye Boulevard, Greenville, North Carolina
  - The Cleveland Clinic Foundation, 9500 Euclid Avenue, Cleveland, Ohio
- Greece (6):
  - University General Hospital of Patras, Department of Internal Medicine, Hematology Division, Rio Patra, Pátrai, Achaia
  - Laiko General Hsoptial of Athens, 16 Sevastoupoleos Street, Athens, Attica
  - University Hospital of Larissa, Mezourlo, Larissa
  - AHEPA University General Hospital of Thessaloniki, Kyriakidi Stilponos 1, Thessaloniki
  - Hippokration Hospital, Konstantinoupoleos 49, Thessaloniki
  - Georgios Papanikolaou General Hospital of Thessaloniki, Exohi, Thessaloniki
- Poland (4):
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Ujejskiego 75, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Smoluchowskiego 17, Gdansk
  - Copernicus PL Sp. z o.o. Wojewodzkie Centrum Onkologii, Aleja Zwyciestwa 31/32, Gdansk
  - EMC Instytut Medyczny S.A Przychondnia przy Łowieckiej, Łowiecka, Wroclaw
- South Korea (5):
  - Ajou University Hospital, 164 World Cup-ro, Yeongtong-gu, Suwon, Gyeonggido
  - Asan Medical Center - PPDS, 88 Olympic-ro 43-gil, Songpa-gu, Seoul
  - Samsung Medical Center PPDS, 81 Irwon-dong Gangnam-gu, Seoul
  - Seoul National University Hospital, 101 Daehak-ro, Jongno-gu, Soeul
  - Severance Hospital Yonsei University Health System, 50-1 Yonsei-Ro, Seodaemun-Gu, Soeul
- Spain (8):
  - Hospital Universitario Quironsalud Madrid, Calle Diego De Velazquez 1, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Ramon y Cajal, Carretera de Colmenar Viejo Km. 9100, Madrid
  - Hospital Universitario 12 de Octubre, Avenida de Cordoba, s/n, Madrid
  - Hospital Universitario La Paz, Paseo Castellana 261, Madrid
  - Hosptial Regional Universitario de Malaga - Hospital General, Avenida Carlos Haya, s/n, Málaga
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Paseo de San Vincent, 58, Salamanca
  - Hospital Universitario Virgen del Rocio, Avenida Manuel Siurot, Centro de Diagnostico y Tratamiento, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Avda Fernando Abril Martorell no° 106, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.fda.gov/Safety/Recalls/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 61 subjects were randomly assigned to receive the study drugs, of whom 60 subjects were included in the ITT set and the safety set each. Note: 1 subject was randomly assigned to the 400 mg BID group but did not receive any dose of study drug as the subject was withdrawn due to noncompliance with the protocol.
Groups:
- SKI-O-703 200 mg BID: 2 capsules of 100 mg SKI-O-703 BID (twice per day)
- SKI-O-703 400 mg BID: 4 capsules of 100 mg SKI-O-703 BID (twice per day)
- Placebo: 4 capsules of placebo BID (twice per day)
Period: Overall Study
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Started | 26 | 22 | 12
Completed | 24 | 20 | 10
Not Completed | 2 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Physician Decision | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo | Total
Number analyzed (Participants) | 26 | 22 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (14.98) | 54.3 (16.3) | 61.1 (22.24) | 56.6 (16.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 5 | 34
  Male | 13 | 6 | 7 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, n(%): Black or African American | 0 | 1 | 0 | 1
  Race, n(%): Asian | 4 | 8 | 1 | 13
  Race, n(%): White | 22 | 13 | 11 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity, n(%): Hispanic or Latino | 2 | 2 | 1 | 5
  Ethnicity, n(%): Not Hispanic or Latino | 24 | 20 | 11 | 55
Number of previous lines of therapy category, n (%) [Count of Participants; unit: Participants]
  0-2 | 9 | 6 | 4 | 19
  ≥3 | 17 | 16 | 8 | 41
Response to previous treatment, n (%) [Count of Participants; unit: Participants]
  Non-responder | 12 | 17 | 9 | 38
  Relapsed | 21 | 18 | 10 | 49
Previous splenectomy, n (%) [Count of Participants; unit: Participants]
  Yes | 6 | 5 | 0 | 11
  No | 20 | 17 | 12 | 49
Baseline platelet count [Mean (Standard Deviation); unit: cells*10^9/L] | 10.6 (6.69) | 11.5 (8.28) | 9.6 (7.22) | 10.7 (7.32)
Baseline platelet count category, n (%) [Count of Participants; unit: Participants]
  <15,000/μL | 19 | 14 | 8 | 41
  15,000/μL-30,000/μL | 7 | 8 | 4 | 19
TPO-receptor agonist use, n (%) [Count of Participants; unit: Participants]
  Yes | 13 | 15 | 7 | 35
  No | 13 | 7 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Platelet Response
Description: Platelet count >= 30,000/µL and doubling the baseline (average of 2 previous counts)
Time Frame: Up to week 12
Population: ITT Set
Measure: Count of Participants; unit: Participants
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
Participants | 12 | 14 | 4

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Discontinuation
Description: The number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs leading to Discontinuation each.
Time Frame: Up to week 16
Measure: Count of Participants; unit: Participants
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
Participants
  Adverse Events (AEs) | 15 | 17 | 8
  Serious Adverse Events (SAEs) | 0 | 2 | 3
  AEs leading to Discontinuation | 2 | 0 | 1

3. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Vital sign measurements considered to be clinically significant in the medical and scientific judgement of the investigator are recorded as AEs.
Time Frame: Up to week 16
Measure: Count of Participants; unit: Participants
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
Participants | 1 | 2 | 0

4. Secondary Outcome: Number of Participants With 12-lead Electrocardiogram (ECG) Abnormalities
Description: 12-lead electrocardiogram (ECG) abnormalities that were recorded as adverse events
Time Frame: Up to week 16
Measure: Count of Participants; unit: Participants
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: Physical examination abnormalities that were recorded as adverse events
Time Frame: Up to week 16
Measure: Count of Participants; unit: Participants
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
Participants | 4 | 4 | 3

6. Secondary Outcome: Quality of Life Score
Description: Qualtiy of Life as measured by the Short Form Questionnaire (SF-36) consists of eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. Scale scores range 0-100 scores (theoritically), with higher scores indicating better health.
  Each health domain score contributes to the Physical Component Summary(PCS) and Mental Component Summary(MCS) scores. Both PCS and MCS are summary scores that are calculated using associated factor weights for the respective summary score applied to all eight scales.
  For overall ranges for PCS and MCS (no theoretical full range available), the SF-36 verion 2 utilizes norm-based scoring involving a linear T-score transformation method so that scores for each of the health domain and component summary measures have a mean of 50 and a standard deviation of 10, based on 2009 U.S. general population. Scores above and below 50 are above and velow the average.
Time Frame: Up to week 16
Population: Safety set defined as all subjects who received at least 1 dose of study drug (SKI-O-703 or placebo).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 23 | 20 | 9
score on a scale
  Physical component summary(Change from baseline) | 0.772 (5.7640) | 0.556 (6.4798) | 1.338 (5.4218)
  Mental component summary(Change from baseline) | 4.913 (11.1022) | -0.930 (8.9426) | 1.643 (10.4183)

7. Secondary Outcome: Consecutive Increased Platelet Counts (≥2 Consecutive PLT ≥ 30,000/µL)
Description: Proportion of participants achieving two or more consecutive platelet counts of ≥ 30,000/μL separated by at least 5 days and without the use of rescue medication
Time Frame: Up to week 12
Population: ITT Set
Measure: Count of Participants; unit: Participants
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
Participants | 10 | 11 | 1

8. Secondary Outcome: Consecutive Increased Platelet Counts (≥2 Consecutive PLT ≥ 50,000/µL)
Description: Proportion of participants achieving two or more consecutive platelet counts of ≥ 50,000/μL separated by at least 5 days and without the use of rescue medication
Time Frame: Up to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
Participants | 5 | 9 | 1

9. Post Hoc Outcome: Bleeding Score
Description: The ITP Bleeding Scale(IBLS) is an immune thrombocytopenic purpura(ITP)-specific bleeding score. The IBLS comprises of 11 site-specific grades, assessed at 9 anatomical sites by history(Hx). In addition, two of these sites, skin and oral, were also assessed by physical examination(PE). These 11 grades include: skin (PE), skin(Hx), oral(PE), oral(Hx), epistaxis, gastrointestinal, urinary, gynecological, pulmonary, intracranial hemorrhage, and subconjunctival hemorrhage, and ranged from Grade 0 (none) to Grade 2 (marked bleeding).
  The grade of IBLS was transformed from categorical type to numerical type (Grade 0 to 0, Grade 1 to 1, Grade 2 to 2, and 0 being better and 2 being worst). Each subject sumed up the transformed scores across all 11 sites per visit assessment. The total overall score ranges from 0-22 with the higher score indicating worst outcome.
Time Frame: Up to week 16
Population: The overall number analyzed is different each visit as patients were dropped.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
Number analyzed (Participants) | 26 | 22 | 12
score on a scale
  Week 1 Day 1: number analyzed (Participants) | 26 | 21 | 12
  Week 1 Day 1 | 2.15 (2.908) | 1.29 (2.411) | 1.75 (2.137)
  Week 5: number analyzed (Participants) | 25 | 21 | 11
  Week 5 | 0.84 (2.249) | 1.33 (3.276) | 0.64 (1.120)
  Week 9: number analyzed (Participants) | 25 | 20 | 11
  Week 9 | 1.16 (3.986) | 0.45 (0.759) | 0.91 (1.640)
  Week 12: number analyzed (Participants) | 24 | 20 | 11
  Week 12 | 1.21 (4.283) | 0.45 (0.759) | 0.55 (1.036)
  End of Study(week 16): number analyzed (Participants) | 24 | 20 | 10
  End of Study(week 16) | 0.42 (0.974) | 0.80 (1.005) | 0.70 (1.160)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: At every study visit, subjects were asked a standard nonleading question to explore a response regarding any medically related changes in their well-being. Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments, including those that worsen from baseline, felt to be clinically significant in the medical and scientific judgment of the investigator were to be recorded as AEs or SAEs.
Arm/Group | SKI-O-703 200 mg BID | SKI-O-703 400 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/22 | 3/12
Other Adverse Events (participants affected / at risk) | 15/26 | 17/22 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SKI-O-703 200 mg BID (N=26) | SKI-O-703 400 mg BID (N=22) | Placebo (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SKI-O-703 200 mg BID (N=26) | SKI-O-703 400 mg BID (N=22) | Placebo (N=12)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 3 (5)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 4 (6) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Corona virus infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT04056195/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04056195/SAP_001.pdf